CLINICAL TRIAL: NCT03810430
Title: Impact of Health Promotion Interventions in Changing Mother's Behavior and Improving Child Health in Hufash District- Al-Mahweet, Yemen
Brief Title: Health Promotion Intervention to Reduce Child Morbidity
Acronym: intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sana'a University (Other)
Responsible Party: Principal Investigator, Mansour Abdu Salah Al-taj, principle investigator, Sana'a University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202016000191-85
Record Dates: First submitted 2019-01-07; First posted 2019-01-18 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Diarrhea; Nutritional
MeSH Terms: conditions — Diarrhea | interventions — Health Promotion

STUDY DESIGN:
Intervention Model Description: The frame work used in this study depends on the Evo-Eco theory of behavior change.This approach consists of five steps; assess, build, create, develop and evaluate (A, B, C, D and E). In the assessment steps, the researcher made a review about the role of water, hygiene and infant feeding promotion in reducing child morbidity and changing mothers' behavior. Based on this review and experience, the researcher developed a baseline questionnaire that was used two months ago before starting the intervention. Based on the results of baseline survey and literature, the researcher with expert team developed the health promotion messages. After developing the messages, interventions took six months. Furthermore, the implementation of the health promotion intervention was at household and community level. Two months later of performing the intervention, the post intervention survey was carried out to measure the primary and secondary outcome of the interventions.
Who Masked: Participant
Masking Description: After baseline survey was carried out, two sub-districts (10 clusters each) were allocated into intervention and control clusters in a 1:1 ratio (10 intervention and 10 control clusters). This allocation of intervention and control clusters was randomly carried out and each sub district had an equal chance of being in either group. For randomization, the two sub districts were listed (1 to 2) and drew randomly by health manager there. Intervention group was informed that participants had been received the intervention, hence it was impossible to fully mask (blind) the study participants. The primary outcomes of interest were measured by observers who were not connected with the intervention implementation, in order to reduce the observer bias
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): ten clusters (villages) were received health promotion activities during six months of interventions
  Interventions: Behavioral: health promotion
- control group (No Intervention): 10 clusters (villages) were not received intervention during the intervention period and by the end of study, it will be compared with the intervention group to measure the change in the primary and secondary outcomes.

INTERVENTIONS:
Behavioral: health promotion — health promotion on water, sanitation and hygiene and child feeding along with hygiene kits were delivered to the mothers in the intervention arm
  Arms: intervention group

SUMMARY:
While household-level water, sanitation and hygiene has been investigated extensively, this is the first comprehensive study to investigate the impact of improved water, sanitation and hygiene and nutrition at household on child health in Yemen.

DETAILED DESCRIPTION:
This study was conducted in Hufash district, Al-Mahweet Province, which is located on the southwest of the capital Sana'a, and takes about (113)kilometers from it. The study aimed to highlight the key role of the community based interventions in reducing child morbidity and mortality in rural Yemen.A community - randomized controlled field trail was implemented to evaluate the role of public health promotion on reducing child diarrhea, acute respiratory infection, nutrition, immunization in children under age of five at enrollment over a six month of study period. Due to the nature of the study, blinding is not possible so some measures would be done to reduce the non-blinding bias like, to keep the study staff blinded as much as possible, the observers and survey staff were not informed about the study design. The sample size required to measure the primary and secondary outcomes before and after the intervention in both groups was estimated using STATA 14.0.Based on data of a previous meta analysis, estimates of required sample size assumed a 20% reduction in the proportion of diarrhea. Intra-cluster correlation coefficient (ICC) was set low at 0.04 and the cluster sizes (number of subjects in a cluster, m) were expected to be 18. The sample size was multiplied by a design effect of 1.68, calculated using DE=1+ICC (m-1), to accommodate the clustering effect. The sample was further adjusted for a potential 20% loss to follow-up over one year, thus requiring a sample of 180 per group. Therefore, the present study estimated that a total of 20 clusters inhabited by 358 households with child aged 6 to 59 months would have 80% power to detect the 20% reduction in the proportion in diarrhea at 5% level of significance.

ELIGIBILITY:
Inclusion Criteria:

* At least one child aged between 6 - 59 months
* Family planning to stay in their home for the next 12 months
* Written consent taken from the head of household

Exclusion Criteria:

* Child had chronic diseases or severely malnourished.
* Family that might leave their house before one year.
* Household that the lord of house refuses to participate.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2015-12-20 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in prevalence of diarrhea among children under five years old | at month 6
  At the end of the six month trial, each household in intervention and control groups are visited by trained field workers to collect morbidity data from mothers or caretakers regarding the daily occurrence of signs and symptoms of child diarrhea. The case definition of diarrhea was 3 or more loose or watery stools over a 24-hour period prior to data collocation.
change in prevalence of acute respiratory infection among children under five years old | at month 6
  At the end of the six month trial, each household in intervention and control groups are visited by trained field workers to collect morbidity data from mothers or caretakers regarding the signs and symptoms of child acute respiratory infection. The case definition of acute respiratory infection was as cough or difficulties with breathing by a child with a raised respiratory rate on two consecutive measurement over a 2 weeks period prior to data collection.
Change in weight-for-age z-score (WAZ) among children age 6 - 59 months | at month 6
  Investigators used 2006 WHO growth reference to calculate WAZ score. Child was considered underweight when child weight for age Z score is below - 2 of the median WHO growth standards
Change in weight-for-height z-score (WHZ) among children age 6 - 59 months | at month 6
  Investigators used 2006 WHO growth reference to calculate WHZ score. Child was considered wasting when child weight for height Z score is below - 2 of the median WHO growth standards
Change in height-for-age z-score (HAZ) among children age 6 - 59 months | at month6
  Investigators used 2006 WHO growth reference to calculate HAZ score. Child was considered stunted when child height for age Z score is below - 2 of the median WHO growth standards

SECONDARY OUTCOMES:
To evaluate the change in mother knowledge about hygiene, water and sanitation as well as child feeding. | at month 6
  Proportion of mothers with improved knowledge regarding water, sanitation and Hygiene as well as child feeding. Face to face interview are conducted with mothers or care givers to measure the level of mother knowledge about water, sanitation and hygiene as well as child feeding.
change in mother hygiene, water and sanitation as well as child feeding behaviors. | at month 6
  Proportion of households with improved water ; proportion of households practicing. To determine water handling practices, hygiene and sanitation practices and child feeding practices, an observation check list is carried out hand washing with soap at the five critical times(before eating, after using latrine, before feeding the child, before cooking and after cleaning child feces); proportion of households disposing of child feces in an improved latrine; proportion of mothers with good child feeding practice.

CONTACTS AND LOCATIONS:
Overall Officials: Abdulwahed A Alserouri, Professor, Principal Investigator — Sanaa University
Locations (1):
- Sanaa University, Sanaa, Yemen

IPD SHARING:
Plan to Share IPD: Undecided
once the results will be ready, we will decide with whom and how can we share the data

REFERENCES:
- [Background] Aiello AE, Coulborn RM, Perez V, Larson EL. Effect of hand hygiene on infectious disease risk in the community setting: a meta-analysis. Am J Public Health. 2008 Aug;98(8):1372-81. doi: 10.2105/AJPH.2007.124610. Epub 2008 Jun 12. PMID 18556606